CLINICAL TRIAL: NCT04622267
Title: Barbed Suture: A Look at Its Use for Hysterotomy Closure During Cesarean Section
Brief Title: Barbed Suture for Hysterotomy Closure During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Calvin Lambert, Assistant Professor-MSH/MSQ/QHC/SSVS/ELM OBGYN FACULTY - ISM, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 20-2571
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Hysterotomy
Keywords: Barbed suture; Blood loss; Hysterotomy; Cesarean section
MeSH Terms: conditions — Hemorrhage | interventions — Polyglactin 910

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the treatment arm or control arm of the study prior to commencement of the cesarean section and following informed consent. Allocation will be concealed to all researchers/providers until this point. The patients will be randomly allocated by block randomization. Generation of random sequence will be done by independent personnel, usually a statistician, who is not going to be involved in the conduct of the RCT. The access to this sequence should be restricted to only a few individuals who absolutely need to have access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard suture (Active Comparator): Standard antimicrobial suture (vicryl) - control arm
  Interventions: Procedure: Standard antimicrobial suture
- Barbed suture (Experimental): Barbed suture type is STRATAFIX Symmetric PDS Plus Knotless Tissue
  Interventions: Device: Barbed suture

INTERVENTIONS:
Device: Barbed suture — to close a C-section incision
  Other Names: STRATAFIX Symmetric PDS Plus Knotless Tissue
  Arms: Barbed suture
Procedure: Standard antimicrobial suture — to close a C-section incision
  Other Names: vicryl
  Arms: Standard suture

SUMMARY:
This is a randomized controlled trial. The purpose of this study is to see if patients whose uterine incision (hysterotomy), at the time of scheduled cesarean section, is closed with barbed suture, have less blood loss compared to women whose incision is closed with the standard suture (vicryl). The primary outcome is quantification of blood loss (QBL). Secondary outcomes include time for hysterotomy closure, need for additional hemostatic sutures, rate of endometritis, use of hemostatic agents, and differences in pain which will be assessed by a telephone screening in the days following delivery.

Study participation will last 1 year and will include the following research procedures :

1. Randomization to barbed suture vs. standard suture
2. Collection of data for primary and secondary outcomes
3. Telephone survey 2 weeks following the procedure to assess pain, bowel/bladder habits, and evidence of wound infection. The barbed suture is approved by the FDA for use in soft tissue approximation and this is not an off-label usage.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial (RCT) evaluating whether using a barbed suture to close a C-section incision can reduce blood loss. Patients undergoing C-section will be randomized with equal allocation to a barbed suture or a standard antimicrobial suture. The primary outcome is quantification of blood loss (QBL). Differences between the groups will be assessed using a 0.05 level Wilcoxon rank-sum test. Secondary outcomes include time for hysterotomy closure, need for additional hemostatic sutures, rate of endometritis/SSI (superficial wound infection, deep wound infection, and endometritis) within 6 weeks postpartum, use of hemostatic agents, and differences in pain which will be assessed by a telephone screening in the days following delivery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a scheduled primary cesarean section at Mount Sinai Hospital
* age 18-64.

Exclusion Criteria:

* Multifetal gestations
* Placenta previas
* Pre-term patients
* Patients with prior uterine incisions or a coagulopathy (DIC, Von Willebrands Disease, etc)
* Patients undergoing an unplanned or emergency cesarean section

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women are the only subjects eligible for this study.
Enrollment: 226 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Lambert, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai Hospital
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfuntner A, Wier LM, Stocks C. Most Frequent Procedures Performed in U.S. Hospitals, 2010. 2013 Feb. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #149. Available from http://www.ncbi.nlm.nih.gov/books/NBK132428/ PMID 23596641
- [Background] Greenberg JA, Goldman RH. Barbed suture: a review of the technology and clinical uses in obstetrics and gynecology. Rev Obstet Gynecol. 2013;6(3-4):107-15. PMID 24920976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment and enrollment conducted from 21 July 2021 through 27 November 2023, and was conducted solely at the Icahn School of Medicine at Mount Sinai Hospital Labor & Delivery Unit at 1176 Fifth Avenue, New York, NY 10029.
Groups:
- Standard Suture: Standard antimicrobial suture (vicryl) to close a C-section incision - control arm
- Barbed Suture: Barbed suture type is STRATAFIX Symmetric PDS Plus Knotless Tissue to close a C-section incision
Period: Overall Study
Arm/Group | Standard Suture | Barbed Suture
Started | 113 | 113
Completed | 113 | 113
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Suture | Barbed Suture | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (5.0) | 35.9 (6.1) | 35.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 113 | 226
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 47
  Not Hispanic or Latino | 88 | 81 | 169
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 57 | 48 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 35 | 62

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Blood Loss
Description: Quantification of blood loss (QBL)
Time Frame: Day 1, At delivery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
mL | 641.8 (300.2) | 596.5 (283.2)

2. Secondary Outcome: Time for Hysterotomy Closure
Description: Time for hysterotomy closure
Time Frame: Day 1, At delivery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
seconds | 326.3 (122.1) | 277.9 (97.3)

3. Secondary Outcome: Number of Participants Who Need Additional Hemostatic Sutures
Time Frame: Day 1, At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
Participants | 50 | 67

4. Secondary Outcome: Number of Hemostatic Sutures
Description: Number of hemostatic sutures needed during procedure
Time Frame: Day 1, At delivery
Measure: Mean (Standard Deviation); unit: sutures
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
sutures | 1.1 (1.2) | 0.9 (1.3)

5. Secondary Outcome: Number of Participants With Surgical Site Infections (SSI)
Description: Number of Participants to assess rate of SSI (any of superficial wound infection, deep wound infection, and endometritis)
Time Frame: Day 1, At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
Participants | 0 | 0

6. Secondary Outcome: Rate of Surgical Site Infections (SSI)
Description: Rate of SSI (any of superficial wound infection, deep wound infection, and endometritis)
Time Frame: 6 weeks
Population: not collected
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Pain Score
Description: Change in pain score at 2 weeks from baseline. Pain score from 0 to 10, with higher score indicating more pain.
  Follow up pain assessment by a telephone screening 2 weeks following delivery.
Time Frame: Day 1, At delivery and 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Suture | Barbed Suture
Number analyzed (Participants) | 113 | 113
score on a scale | 3.1 (1.0) | 3.1 (1.0)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Standard Suture | Barbed Suture
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 1/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Suture (N=113) | Barbed Suture (N=113)
intrapartum hematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04622267/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT04622267/ICF_001.pdf